CLINICAL TRIAL: NCT04977011
Title: Effectiveness of Music Intervention on Anxiety in Critical Ill Patient: Randomized Controlled Trial
Brief Title: Effectiveness of Music Intervention on Anxiety and Physiological Responses in Critical Ill Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MSIRB2018020
Record Dates: First submitted 2021-07-05; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Ketoacidosis; Heart Disease, Ischemic; Stroke; GastroIntestinal Bleeding; Acute Kidney Injury; Heart Failure; Trauma; Septic Shock; Respiratory Failure; Pneumonia; Intracerebral Hemorrhage; Head Injury; Liver Diseases
Keywords: Music intervention; Anxiety; Agitation; Sleep quality; Intensive Care Unit
MeSH Terms: conditions — Diabetic Ketoacidosis; Myocardial Ischemia; Stroke; Gastrointestinal Hemorrhage; Acute Kidney Injury; Heart Failure; Wounds and Injuries; Shock, Septic; Respiratory Insufficiency; Pneumonia; Cerebral Hemorrhage; Craniocerebral Trauma; Liver Diseases; Anxiety Disorders; Psychomotor Agitation; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: 30 minutes music intervention for 3 days on bedside
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 30 minutes music intervention for 3 days on bedside
  Interventions: Other: relaxing music
- control group (No Intervention): usually care

INTERVENTIONS:
Other: relaxing music — 30 minutes relaxing music for continuity 3 days since admission
  Arms: experimental group

SUMMARY:
Music intervention is a non-pharmacological and effective intervention that can alleviate anxiety and agitation in patients undergoing weaning. The effectiveness of music intervention in reducing anxiety of patients in Intensive Care Unit (ICU) is still unknown. The purpose of this study was to examine the effectiveness of music intervention on anxiety, agitation, sleep quality and physiological parameters on patients in ICU. This study was conducted from January to June 2019. A total of 196 hospitalized ICU patients were divided into two groups. Subjects in experimental group received 30 minutes music intervention for 3 days on bedside whereas subjects in control group received routine care only. The primary outcome was anxiety. Agitation Sedation Scale, sleep quality and physical parameters were selected to collect as secondary outcomes.There was no significant difference between the groups at baseline. The results of this study support that music can reduce anxiety and agitation levels in ICU's patient. Nurses can incorporate this intervention into the daily care in order to reduce the discomfort of patients.

DETAILED DESCRIPTION:
Background:Music intervention is a non-pharmacological and effective intervention that can alleviate anxiety and agitation in patients undergoing weaning. The effectiveness of music intervention in reducing anxiety of patients in ICU is still unknown.

Objectives: The purpose of this study was to examine the effectiveness of music intervention on anxiety, agitation, sleep quality and physiological parameters on patients in ICU.

Methods: This study was conducted from January to June 2019. A total of 196 hospitalized ICU patients were divided into two groups. Subjects in experimental group received 30 minutes music intervention for 3 days on bedside whereas subjects in control group received routine care only. The primary outcome was anxiety measured by Visual Analog Scale. Richmond Agitation Sedation Scale, Richards-Campbell Sleep Scale and their physical parameters were selected to collect the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or older and staying in an intensive care unit.
* Patients within 24 hours of admission (Acute Physiology And Chronic Health Evaluation, APACHE II score) ≦25 points.
* Can express their intentions by writing or shaking their heads.
* Can communicate in Mandarin, Taiwanese, Hakka or English.
* After explaining the purpose of the research, agree to participate and fill out the consent form.

Exclusion Criteria:

* Dementia or mental illness are recorded

Ages: 20 Years to 102 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Anxiety Visual Analog Scale. | 3day
  The Visual Analogue Scale for Anxiety (VASA) is a line 10 centimetres in length with "not at all anxious" and "very anxious" at the left and right extremes respectively.

SECONDARY OUTCOMES:
Richmond Agitation Sedation Scale | 3 day
  The Richmond Agitation-Sedation Scale (RASS) was developed in a collaborative effort with practitioners representing critical care physicians, nurses, and pharmacists. RASS is a 10-point scale, with four levels of anxiety or agitation (+1 to +4 [combative]), one level to denote a calm and alert state (0), and 5 levels of sedation (-1 to -5) culminating in unarousable (-5).
Richards-Campbell Sleep Scale | 3 day
  The RCSQ is used in order to assess sleep quality in eligible ICU patients. The RCSQ is a six-item self-report questionnaire that is used in order to assess perceived sleep depth, sleep latency (time to fall asleep), and number of awakenings, as well as sleep efficiency, quality and perceived nighttime noise. Each RCSQ item is scored on a visual analog scale ranging from 0 mm to 100 mm, with higher scores representing better sleep. The mean score of the six items is known as the total score and represents the overall perception of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Han Tsai, Study Chair — Min-Sheng General Hospital
Locations (1):
- MinSheng General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aghaie B, Rejeh N, Heravi-Karimooi M, Ebadi A, Moradian ST, Vaismoradi M, Jasper M. Effect of nature-based sound therapy on agitation and anxiety in coronary artery bypass graft patients during the weaning of mechanical ventilation: A randomised clinical trial. Int J Nurs Stud. 2014 Apr;51(4):526-38. doi: 10.1016/j.ijnurstu.2013.08.003. Epub 2013 Aug 29. PMID 24035670
- [Result] Chlan LL, Weinert CR, Heiderscheit A, Tracy MF, Skaar DJ, Guttormson JL, Savik K. Effects of patient-directed music intervention on anxiety and sedative exposure in critically ill patients receiving mechanical ventilatory support: a randomized clinical trial. JAMA. 2013 Jun 12;309(22):2335-44. doi: 10.1001/jama.2013.5670. PMID 23689789
- [Result] Cook D, Rocker G. Dying with dignity in the intensive care unit. N Engl J Med. 2014 Jun 26;370(26):2506-14. doi: 10.1056/NEJMra1208795. No abstract available. PMID 24963569
- [Result] Dijkstra BM, Gamel C, van der Bijl JJ, Bots ML, Kesecioglu J. The effects of music on physiological responses and sedation scores in sedated, mechanically ventilated patients. J Clin Nurs. 2010 Apr;19(7-8):1030-9. doi: 10.1111/j.1365-2702.2009.02968.x. PMID 20492047
- [Result] Golino AJ, Leone R, Gollenberg A, Christopher C, Stanger D, Davis TM, Meadows A, Zhang Z, Friesen MA. Impact of an Active Music Therapy Intervention on Intensive Care Patients. Am J Crit Care. 2019 Jan;28(1):48-55. doi: 10.4037/ajcc2019792. PMID 30600227
- [Result] Han L, Li JP, Sit JW, Chung L, Jiao ZY, Ma WG. Effects of music intervention on physiological stress response and anxiety level of mechanically ventilated patients in China: a randomised controlled trial. J Clin Nurs. 2010 Apr;19(7-8):978-87. doi: 10.1111/j.1365-2702.2009.02845.x. PMID 20492042
- [Result] Johnson K, Fleury J, McClain D. Music intervention to prevent delirium among older patients admitted to a trauma intensive care unit and a trauma orthopaedic unit. Intensive Crit Care Nurs. 2018 Aug;47:7-14. doi: 10.1016/j.iccn.2018.03.007. Epub 2018 May 4. PMID 29735284
- [Result] Korhan EA, Khorshid L, Uyar M. The effect of music therapy on physiological signs of anxiety in patients receiving mechanical ventilatory support. J Clin Nurs. 2011 Apr;20(7-8):1026-34. doi: 10.1111/j.1365-2702.2010.03434.x. Epub 2011 Feb 16. PMID 21323778
- [Result] Lee OK, Chung YF, Chan MF, Chan WM. Music and its effect on the physiological responses and anxiety levels of patients receiving mechanical ventilation: a pilot study. J Clin Nurs. 2005 May;14(5):609-20. doi: 10.1111/j.1365-2702.2004.01103.x. PMID 15840076
- [Result] Lee WP, Wu PY, Lee MY, Ho LH, Shih WM. Music listening alleviates anxiety and physiological responses in patients receiving spinal anesthesia. Complement Ther Med. 2017 Apr;31:8-13. doi: 10.1016/j.ctim.2016.12.006. Epub 2017 Jan 7. PMID 28434475
- [Result] Liang Z, Ren D, Choi J, Happ MB, Hravnak M, Hoffman LA. Music intervention during daily weaning trials-A 6 day prospective randomized crossover trial. Complement Ther Med. 2016 Dec;29:72-77. doi: 10.1016/j.ctim.2016.09.003. Epub 2016 Sep 15. PMID 27912960
- [Result] Najafi Ghezeljeh T, Mohaddes Ardebili F. Comparing the effect of patients preferred music and Swedish massage on anticipatory anxiety in patients with burn injury: Randomized controlled clinical trial. Complement Ther Clin Pract. 2018 Aug;32:55-60. doi: 10.1016/j.ctcp.2018.05.002. Epub 2018 May 4. PMID 30057058
- [Result] Papathanassoglou EDE, Hadjibalassi M, Miltiadous P, Lambrinou E, Papastavrou E, Paikousis L, Kyprianou T. Effects of an Integrative Nursing Intervention on Pain in Critically Ill Patients: A Pilot Clinical Trial. Am J Crit Care. 2018 May;27(3):172-185. doi: 10.4037/ajcc2018271. PMID 29716903
- [Result] Phipps MA, Carroll DL, Tsiantoulas A. Music as a therapeutic intervention on an inpatient neuroscience unit. Complement Ther Clin Pract. 2010 Aug;16(3):138-142. doi: 10.1016/j.ctcp.2009.12.001. Epub 2010 May 15. PMID 20621273
- [Result] Saadatmand V, Rejeh N, Heravi-Karimooi M, Tadrisi SD, Zayeri F, Vaismoradi M, Jasper M. Effect of nature-based sounds' intervention on agitation, anxiety, and stress in patients under mechanical ventilator support: a randomised controlled trial. Int J Nurs Stud. 2013 Jul;50(7):895-904. doi: 10.1016/j.ijnurstu.2012.11.018. Epub 2012 Dec 14. PMID 23245705
- [Result] Su CP, Lai HL, Chang ET, Yiin LM, Perng SJ, Chen PW. A randomized controlled trial of the effects of listening to non-commercial music on quality of nocturnal sleep and relaxation indices in patients in medical intensive care unit. J Adv Nurs. 2013 Jun;69(6):1377-89. doi: 10.1111/j.1365-2648.2012.06130.x. Epub 2012 Aug 29. PMID 22931483
- [Result] Wong HL, Lopez-Nahas V, Molassiotis A. Effects of music therapy on anxiety in ventilator-dependent patients. Heart Lung. 2001 Sep-Oct;30(5):376-87. doi: 10.1067/mhl.2001.118302. PMID 11604980